CLINICAL TRIAL: NCT05312190
Title: Clinical and Basic Researches Related to ZhenQi Buxue Oral Liquid in Treating Menstrual Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: West China Second University Hospital (Other); Chongqing Medical University No.1 Affiliated Hospital (Unknown); The Second Hospital of Hebei Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); Zhongda Hospital (Other); Hubei Maternal and Child Health Hospital (Unknown); Liuzhou Maternity and Child Healthcare Hospital (Other); Zhejiang University Medical College Affiliated Hangzhou First People's Hospital (Unknown); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZhenQi202201
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Menstrual Disorders
Keywords: Menstrual disorders; Traditional Chinese medicine
MeSH Terms: conditions — Menstruation Disturbances | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: This study is a national multicenter prospective, randomized, controlled trial. One third of participanta will receive Zhenqi Buxue Oral Liquid, one third of participanta will receive Progesterone Capsules, and the another third will receive Zhenqi Buxue Oral Liquid and Progesterone Capsules in combination.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zhenqi Buxue Oral Liquid (Experimental): Zhenqi Buxue Oral Liquid, 10 ml each time, 2 times a day for 3 menstrual cycles, orally
  Interventions: Drug: ZhenQi BuXue KouFuYe
- Zhenqi Buxue Oral Liquid and Progesterone Capsules (Experimental): Zhenqi Buxue Oral Liquid was taken orally, 10 ml at a time, twice a day for 3 menstrual cycles + orally from the second half of menstrual cycle, Progesterone Capsules 200mg, once a day for 10 days for 3 menstrual cycles
  Interventions: Drug: ZhenQi BuXue KouFuYe; Drug: Progesterone Capsules
- Progesterone Capsules (Active Comparator): Progesterone Capsules 200mg, qd*10 days*3 menstrual cycles, orally
  Interventions: Drug: Progesterone Capsules

INTERVENTIONS:
Drug: ZhenQi BuXue KouFuYe — Zhenqi Buxue Oral Liquid consists of sheep placenta, pearl, red ginseng, wolfberry, astragalus, angelica, coix seed, ginger and jujube. The excipients are protein sugar and sodium benzoate. Nourishes qi and blood. It is suitable for dizziness, pale complexion, fatigue, lack of energy and lazy words caused by insufficient qi and blood.
  Arms: Zhenqi Buxue Oral Liquid; Zhenqi Buxue Oral Liquid and Progesterone Capsules
Drug: Progesterone Capsules — The main ingredient of Progesterone Capsules is abbsolutely progesterone,a kind of hormone,which is the main method of western medicine for the treatment of menstrual disorders
  Arms: Progesterone Capsules; Zhenqi Buxue Oral Liquid and Progesterone Capsules

SUMMARY:
This study is a national multicenter prospective, randomized, controlled trial, which evaluates Zhenqi Buxue Oral Liquid，Progesterone Capsules and the addition of Zhenqi Buxue Oral Liquid to Progesterone Capsules in the treatment of menstrual disorders in adults women. One third of participanta will receive Zhenqi Buxue Oral Liquid, one third of participanta will receive Progesterone Capsules, and the another third will receive Zhenqi Buxue Oral Liquid and Progesterone Capsules in combination.

DETAILED DESCRIPTION:
Menstrual disorders are one of the most common clinical symptoms in women. Since puberty, about 70% of women have experienced menstrual disorders, including early, delayed, shortened, prolonged, and more importantly oligomenorrhea, amenorrhea, and decreased menstrual flow.At present, the main method of western medicine for the treatment of menstrual disorders is hormone replacement therapy, but the incidence of adverse reactions is high, and the clinical effect is mediocre. Traditional Chinese medicine in my country mostly adopts holistic conditioning therapy for the treatment of irregular menstruation.

Zhenqi Buxue Oral Liquid consists of sheep placenta, pearl, red ginseng, wolfberry, astragalus, angelica, coix seed, ginger and jujube. The excipients are protein sugar and sodium benzoate. Nourishes qi and blood. It is suitable for dizziness, pale complexion, fatigue, lack of energy and lazy words caused by insufficient qi and blood.

This study will conduct a comprehensive and in-depth study on its treatment of mental and psychological stress and menstrual disorders with "oligomenorrhea, amenorrhea, amenorrhea and decreased menstrual flow" as the main manifestations. The molecular mechanism and clinical improvement, and the safety and adverse reactions of its use paln to be clarified.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 25 and 40 years old;
2. Patients with oligomenorrhea or oligomenorrhea or menopause within three months (see Appendix 1: Diagnostic Criteria of Traditional Chinese and Western Medicine)
3. Meet the clinical medication conditions for progesterone to regulate menstruation
4. The research subjects were informed and voluntarily participated in this study, and signed the informed consent at the same time.

Exclusion Criteria:

1. Age <25 years or >40 years old, pregnant or breastfeeding women
2. Ovarian dysfunction caused by local ovarian surgery, radiotherapy and chemotherapy for previous malignant tumors, taking hormones or immunosuppressive drugs;
3. Combined with serious or unstable physical diseases that may affect the efficacy of drugs and the conduct of trials, including liver, kidney, gastrointestinal, cardiovascular, respiratory, endocrine, neurological, immune or blood system diseases, etc., mental patients .
4. Those who were allergic to the drugs used in the trial or had serious adverse reactions in the past;
5. Breast cancer or family history of breast cancer in first-degree relatives, irregular vaginal bleeding, uterine fibroids (≥3cm), endometriosis, atypical endometrial hyperplasia, endometrial cancer and other hormone-dependent reproduction Systemic diseases and other malignant tumors;
6. Those with a history of thromboembolic disease or thrombosis;
7. Participated in a clinical trial of another research drug within 3 months prior to inclusion in this study (the first interview);
8. Those who have used related drugs in the past 3 months or have abused or depended on substances (alcohol or drugs) in the past 3 months; heavy smokers (smokers who smoke 20 or more cigarettes per day);
9. Those who met the inclusion criteria, did not follow the doctor's advice, were unable to judge the curative effect or were unable to evaluate the curative effect due to incomplete data.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 330 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual improvement | Within 3 months after the trial complete
  Menstrual improvement in cycle period
Menstrual improvement | Within 3 months after the trial complete
  Menstrual improvement in menstrual volume
Menstrual improvement | Within 3 months after the trial complete
  Menstrual improvement in number of days with bleeding or spotting
Menstrual improvement | Within 3 months after the trial complete
  Menstrual improvement in monthly rates of amenorrhea

SECONDARY OUTCOMES:
Sex hormone levels | Within 3 months after the trial complete
  mainly FSH, LH，E2 and AMH
AFC | Within 3 months after the trial complete
  Changes in AFC in pelvic ultrasonography
SF-36 | Within 3 months after the trial complete
  The change of the MOS item short from health survey

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Lei Li, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05312190/Prot_SAP_ICF_000.pdf